CLINICAL TRIAL: NCT05556096
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel, Multicenter Study to Evaluate the Safety and Efficacy of ALXN1720 in Adults With Generalized Myasthenia Gravis
Brief Title: Safety and Efficacy of ALXN1720 in Adults With Generalized Myasthenia Gravis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALXN1720-MG-301; 2022-000460-21 (EudraCT Number)
Record Dates: First submitted 2022-09-23; First posted 2022-09-27 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Generalized Myasthenia Gravis
Keywords: ALXN1720; anti-acetylcholine receptor antibody-positive; acetylcholine receptor; AChR; generalized myasthenia gravis; myasthenia gravis; MG; gMG; complement component 5; C5; VHH antibody
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Intervention Model Description: This is a treatment study with 2 parallel intervention groups. The study is blinded for sponsor staff, sponsor designees, investigative site personnel, other staff directly associated with the conduct of the study, and study participants.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- ALXN1720 (Experimental): Participants will receive a weight-based initial (loading) dose of ALXN1720 on Day 1, followed by weight-based maintenance treatment with ALXN1720 on Day 8 and once every week (Q1W) thereafter for a total of 26 weeks. Following this randomized controlled treatment (RCT) period, all participants will receive ALXN1720 in an open-label extension (OLE) period of 105 weeks.
  Interventions: Combination Product: ALXN1720
- Placebo (Placebo Comparator): Participants will receive placebo during the 26-week RCT period, after which they will enter the OLE period of the study and receive ALXN1720.
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: ALXN1720 — Combination product consisting of syringe prefilled with ALXN1720.
  Arms: ALXN1720
Combination Product: Placebo — Combination product consisting of syringe prefilled with placebo.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ALXN1720 for the treatment of generalized MG (gMG) in adults with autoantibodies against acetylcholine receptor (AChR).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MG with generalized muscle weakness meeting the clinical criteria defined by Myasthenia Gravis Foundation of America (MGFA) Class II, III or IV
* Positive serological test for autoantibodies against AChR

Exclusion Criteria:

* History of thymectomy, or any other thymic surgery within 12 months prior to Screening
* Untreated thymic malignancy, carcinoma, or thymoma
* History of Neisseria meningitidis infection
* Pregnancy, breastfeeding, or intention to conceive during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Myasthenia Gravis-Activities of Daily Living (MG-ADL) Total Score at Week 26 | Baseline, Week 26

SECONDARY OUTCOMES:
Change From Baseline in Quantitative Myasthenia Gravis (QMG) Total Score at Week 26 | Baseline, Week 26
Percentage of Responders Based on Reduction of the MG-ADL Total Score at Week 26 | Baseline up to Week 26
  Response is defined as reduction of the MG-ADL total score by >= 3 points from baseline at Week 26.
Percentage of Responders based on Reduction of the QMG Total Score at Week 26 | Baseline up to Week 26
  Response is defined as reduction of the QMG total score by >= 5 points from baseline at Week 26
Change From Baseline in Myasthenia Gravis Composite (MGC) Total Score at Week 26 | Baseline, Week 26
Change from Baseline in the QMG total score at Week 4 | Baseline, Week 4

CONTACTS AND LOCATIONS:
Locations (118):
- United States (23):
  - Research Site, Orange, California
  - Research Site, Fort Collins, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Bradenton, Florida
  - Research Site, Maitland, Florida
  - Research Site, Tampa, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Gainesville, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Springfield, Illinois
  - Research Site, Kansas City, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Detroit, Michigan
  - Research Site, East Lansing, Michigan
  - Research Site, Las Vegas, Nevada
  - Research Site, Patchogue, New York
  - Research Site, Rochester, New York
  - Research Site, Syracuse, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, North Charleston, South Carolina
  - Research Site, Houston, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Morgantown, West Virginia
- Argentina (3):
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Rosario
- Austria (2):
  - Research Site, Innsbruck
  - Research Site, Wels
- Brazil (7):
  - Research Site, Barretos
  - Research Site, Joinville
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, Salvador
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Canada (3):
  - Research Site, Edmonton, Alberta
  - Research Site, Toronto, Ontario
  - Research Site, Québec, Quebec
- China (12):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Fuzhou
  - Research Site, Hangzhou
  - Research Site, Jinan
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Suzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
- Denmark (2):
  - Research Site, Aalborg
  - Research Site, Copenhagen
- France (6):
  - Research Site, Garches
  - Research Site, Lille
  - Research Site, Marseille
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Strasbourg
- Germany (4):
  - Research Site, Berlin
  - Research Site, Düsseldorf
  - Research Site, München
  - Research Site, Würzburg
- Israel (3):
  - Research Site, Hadera
  - Research Site, Haifa
  - Research Site, Petah Tikva
- Italy (9):
  - Research Site, Bergamo
  - Research Site, Brescia
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Palermo
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Rome
- Japan (11):
  - Research Site, Chiba
  - Research Site, Fukushima
  - Research Site, Higashimatsuyama-shi
  - Research Site, Isehara-shi
  - Research Site, Itabashi-ku
  - Research Site, Kawasaki-shi
  - Research Site, Morioka
  - Research Site, Nagasaki
  - Research Site, Nagoya
  - Research Site, Shinjuku-ku
  - Research Site, Suita-shi
- Research Site, Amsterdam, Netherlands
- Poland (5):
  - Research Site, Bydgoszcz
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Poznan
- Portugal (2):
  - Research Site, Almada
  - Research Site, Porto
- Serbia (2):
  - Research Site, Belgrade
  - Research Site, Niš
- South Korea (4):
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Gwangju
  - Research Site, Seoul
- Spain (6):
  - Research Site, Badalona (Barcelona)
  - Research Site, Córdoba
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Seville
- Research Site, Sankt Gallen, Switzerland
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Tainan
  - Research Site, Taipei
- Turkey (Türkiye) (4):
  - Research Site, Bursa
  - Research Site, Istanbul
  - Research Site, Kocaeli
  - Research Site, Samsun
- United Kingdom (4):
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Oxford
  - Research Site, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.